CLINICAL TRIAL: NCT06563869
Title: Efficacy and Safety of Sintilimab in Combination With Platinum-containing Chemotherapy Plus PEG-rhG-GSF for Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma: a Prospective, Open, Single-arm, Single-center Clinical Study
Brief Title: Sintilimab With Chemotherapy Plus PEG-rhG-GSF for Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 12
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma, PEG-rhG-GSF
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Intervention Model Description: All subjects who meet the inclusion criteria will receive sintilimab combined with platinum-containing chemotherapy for 2 cycles (21 days for 1 cycle) as neoadjuvant therapy according to the research plan. Polyethylene glycolylated recombinant human granulocyte stimulating factor will be given 24 hours after the end of chemotherapy. Radical surgical treatment will be received within 3-6 weeks after the completion of the last neoadjuvant treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant patients (Experimental): All subjects who meet the inclusion criteria will receive sintilimab combined with platinum-containing chemotherapy for 2 cycles (21 days for one cycle) as neoadjuvant therapy according to the research plan. Polyethylene glycolylated recombinant human granulocyte stimulating factor will be given 24 hours after the end of chemotherapy. Radical surgical treatment will be received within 3 to 6 weeks after the completion of the last neoadjuvant treatment.
  Interventions: Drug: PEG-rhG-GSF

INTERVENTIONS:
Drug: PEG-rhG-GSF — Polyethylene glycolylated recombinant human granulocyte stimulating factor （6mg）will be given 24 hours after the end of chemotherapy.
  Other Names: Polyethylene glycolylated recombinant human granulocyte stimulating factor

SUMMARY:
This study is a prospective, open-label, single-arm, single-center clinical study, aiming to evaluate the efficacy and safety of sintilimab combined with platinum-based chemotherapy + pegylated recombinant human granulocyte stimulating factor as neoadjuvant treatment for resectable esophageal squamous cell carcinoma patients. In the study, all patients who meet the inclusion criteria will receive sintilimab combined with platinum-based chemotherapy for 2 cycles (21 days as one cycle) as neoadjuvant treatment according to the study plan. Pegylated recombinant human granulocyte stimulating factor will be given 24 hours after the end of chemotherapy, and radical surgical treatment will be received within 3-6 weeks after the completion of the last neoadjuvant treatment. Whether the subjects need adjuvant treatment after surgery and the adjuvant treatment plan will be determined by the investigators. All subjects need to complete the follow-up plan formulated by the study after surgery.

DETAILED DESCRIPTION:
The patients selected for the study were those who were diagnosed with esophageal cancer for the first time. The recruited subjects should be:

1. Preoperatively, the main part of the tumor was located in the middle and lower part of the esophagus (below 18 cm from the incisors) as shown by gastroscopy, and the pathological type was squamous cell carcinoma as shown by biopsy.
2. Preoperatively, patients with esophageal cancer assessed by imaging (CT, MRI or PET/CT), cervical B-ultrasound and endoscopic ultrasound as potentially resectable. Potentially resectable patients were defined as those with T2-4aNxM0, stage II-IVA (AJCC staging, 8th edition, 2017) of esophageal cancer according to the 2022 Guidelines for the Diagnosis and Treatment of Esophageal Cancer of the Chinese Society of Clinical Oncology. For T2N0M0, the length of the primary tumor under endoscopic examination was required to be ≥ 2 cm, located below the neck, and ≥ 5 cm away from the cricopharyngeal muscle.
3. Signed the informed consent form and met all the inclusion and exclusion criteria of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent;
2. Male or female, aged 18 years or above and 75 years or below;
3. Patients diagnosed with esophageal squamous cell carcinoma by biopsy histopathological examination of the primary lesion; cervical metastasis was excluded by cervical B-ultrasound.
4. Patients who were judged by imaging and endoscopic ultrasound examination to have potentially surgically resectable middle and lower esophagus (below 18 cm from the incisors) and require neoadjuvant therapy (T2-4aNxM0, stage II-IVA); for T2N0M0, the length of the primary tumor under endoscopic examination was required to be ≥ 2 cm, located below the neck, and ≥ 5 cm away from the cricopharyngeal muscle.
5. Patients have not received any anti-tumor treatment in the past, including but not limited to surgery, radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc.;
6. The ECOG performance status score is 0-1;
7. Have adequate heart, lung, liver and kidney functions, and the laboratory tests within 14 days before screening meet the following indicators:

   i. Hemoglobin HB ≥ 90 g/L ii. Absolute neutrophil count ANC ≥ 1.5 × 109 /L iii. Platelet count PLT ≥ 80 × 109 /L iv. Albumin ALB ≥ 35 g/L v. Alanine aminotransferase ALT and aspartate aminotransferase AST ≤ 1.5 times the upper limit of the normal range vi. Total bilirubin ≤ 30 μmol/L vii. Creatinine SCr ≤ the upper limit of the normal range. viii. Coagulation: PT-INR ≤ 2.3 or PT < 6 seconds compared with the normal control
8. Patients need to be able to complete the treatment and follow-up according to the research plan on schedule;
9. Patients need to have sufficient tissue samples and agree to use their tissue samples and blood samples for research analysis;
10. Pregnancy tests in women of childbearing age were negative and were willing to take effective contraceptive measures during the study.

Exclusion Criteria:

1. Patients who may have tracheoesophageal fistula or aortic esophageal fistula;
2. Patients with severe malnutrition or in need of tube feeding;
3. Patients with other malignant tumors within 2 years and not cured (except for cured basal cell carcinoma of the skin and cervical carcinoma in situ);
4. Patients with active autoimmune system diseases, or with a history of autoimmune system diseases or symptoms and in need of systemic hormone therapy or anti-autoimmune drug therapy;
5. Patients with immunodeficiency, or still receiving systemic steroid hormone therapy (prednisone > 10 mg/day or other equivalent drugs) 7 days before the administration of the first dose of neoadjuvant therapy in this study, or other forms of immunosuppressive therapy;
6. Patients with active infection and still in need of systemic treatment 7 days before the administration of the first dose of neoadjuvant therapy in this study;
7. Patients with uncontrollable systemic diabetes;
8. Patients with interstitial lung disease, non-infectious pneumonia or pulmonary fibrosis;
9. Patients with previous motor nerve or sensory nerve toxicity symptoms greater than WHO grade 1;
10. Patients who have received allogeneic organ or stem cell transplantation in the past;
11. Patients allergic to the drugs or related components involved in this study;
12. Patients currently participating in other clinical studies;
13. Patients who received anti-programmed death-1 (PD-1)/PD-1 ligand (PD-L1) monoclonal antibodies, cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibodies or other immune or molecular targeted therapies within 4 weeks before screening;
14. Patients with any serious or unstable medical conditions or mental illnesses;
15. Patients with known active alcohol or drug abuse or dependence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
pCR | Radical surgical treatment will be received within 3 to 6 weeks after the completion of the last neoadjuvant treatment.
  The pathological complete response rate (pCR) after neoadjuvant therapy

SECONDARY OUTCOMES:
MPR | Radical surgical treatment will be received within 3 to 6 weeks after the completion of the last neoadjuvant treatment.
  major pathological response, MPR
RFS | 5 years
  Recurrence Free Survival
R0 resection rate | Radical surgical treatment will be received within 3 to 6 weeks after the completion of the last neoadjuvant treatment.
  The R0 resection rate after neoadjuvant therapy and subsequent surgery
AEs | 4 years
  New adjuvant therapy-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Gu, Ph.D., Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No